CLINICAL TRIAL: NCT05024708
Title: Athlete's Heart or Arrhythmogenic Right Ventricular Cardiomyopathy: Contribution of Exercise Cardiovascular Magnetic Resonance (CMR)
Acronym: CA2VD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 35RC21_9886_CA2VD
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Arrhythmogenic Right Ventricular Cardiomyopathy
Keywords: ARVC, Athlete's heart, exercise, CMR, RV contractile reserve
MeSH Terms: conditions — Arrhythmogenic Right Ventricular Dysplasia; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ARVC patients (Experimental)
  Interventions: Other: Cardiac exercises and tests
- Endurance athletes with a dilated RV (Active Comparator)
  Interventions: Other: Cardiac exercises and tests
- Endurance athletes with normal RV (Active Comparator)
  Interventions: Other: Cardiac exercises and tests
- Untrained subject with normal RV (Experimental)
  Interventions: Other: Cardiac exercises and tests

INTERVENTIONS:
Other: Cardiac exercises and tests — Rest ECG, rest echocardiography, cardio-pulmonary exercise test, exercise echocardiography, holter ECG monitor (48 yours), rest CMR, exercise CMR (ergocycle)

SUMMARY:
Prospective, nonrandomized, single-center, comparative study to define if right ventricular (RV) contractile reserve assessed by exercise CMR helps to improve the differential diagnosis between pathological and physiological remodeling of the RV; ie. arrhythmogenic right ventricular cardiomyopathy (ARVC) and athlete's heart.

DETAILED DESCRIPTION:
Comparison of the RV contractile reserve in 4 groups of patients: Arrhythmogenic right ventricular cardiomyopathy (ARVC) patients; endurance athletes with a dilated RV, endurance athletes with normal RV, untrained subject with normal RV.

Patients will come to the hospital for 3 visits (3 half days):

* Visit 1: clinical evaluation, rest ECG, rest echocardiography, cardio-pulmonary exercise test.
* Visit 2: exercise echocardiography, holter ECG monitor (48 yours)
* Visit 3: rest CMR and exercise CMR (ergocycle)

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 years and older,

  * patients with confirmed ARVC, but with no major RV dysfunction (RVEF >40%)
  * endurance athletes with dilated RV
  * endurance athletes with non-dilated RV
  * untrained healthy subjects with non-dilated RV
* who signed a written free and informed consent:

Exclusion Criteria:

* Patients with other cardiovascular disease;
* Contra-indication to CMR (in particular presence of a non-CMR compatible implantable cardiac defibrillator);
* Patients with permanent supraventricular arrhythmia;
* Patients unable to perform an exercise test on an ergocycle;
* Person subject to legal protection (safeguard justice, trusteeship and guardianship) and persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2024-01-16 (Estimated); Study Completion 2024-01-16 (Estimated)

PRIMARY OUTCOMES:
Evolution of right ventricular ejection fraction (RVEF) assessed with CMR during exercise | Through study completion, an average of 1 month

SECONDARY OUTCOMES:
Evolution of Tricuspid annular plane systolic excursion (TAPSE) during exercise | Through study completion, an average of 1 month
Evolution of S' tricuspid wave during exercise | Through study completion, an average of 1 month
Evolution of RV fractional area during exercise | Through study completion, an average of 1 month
Evolution of free wall RV strain during exercise | Through study completion, an average of 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No